CLINICAL TRIAL: NCT06275750
Title: Non-surgical Spinal Decompression in Patients With Chronic Low Back Pain and Sciatica: a 2-month Follow-up Study
Brief Title: Non-surgical Spinal Decompression in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Armando Tonatiuh Avila Garcia, Chief Department of Physical Medicine and Rehabilitation, Hospital Civil de Guadalajara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEI 175/23
Record Dates: First submitted 2024-02-09; First posted 2024-02-23 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain; Sciatica; Lumbar Disc Herniation
MeSH Terms: conditions — Low Back Pain; Sciatica; Intervertebral Disc Displacement | interventions — Laminectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients treated with non-surgical spinal decompression (Experimental): The patients were positioned in supine with adjustable lumbar, and thoracic belts attached to the traction cord. After tightening the belts, the M7 position was selected to achieve hip and knee flexion, and posterior pelvic tilt of 25° was added. Before starting the therapy, the weight of the subject was entered in the panel, and a short tolerance test was carried out. Patients were provided with a manual switch to stop treatment any time. Preset lumbar disc herniation protocol was used. Each session lasted fifteen minutes, applied force had 100-gram step increments, and did not exceed 50% of the weight of the patient. At the end of the therapy, the cord was disconnected and belts were removed. Participants were asked to sit for three minutes to identify any adverse reaction.
  Interventions: Device: Spinal decompression with BTL-6000 spinal decompression system (BTL Industries Ltd.)

INTERVENTIONS:
Device: Spinal decompression with BTL-6000 spinal decompression system (BTL Industries Ltd.) — The patients were positioned in supine with adjustable lumbar, and thoracic belts attached to the traction cord. After tightening the belts, the M7 position was selected to achieve hip and knee flexion, and posterior pelvic tilt of 25° was added. Before starting the therapy, the weight of the subject was entered in the panel, and a short tolerance test was carried out. Patients were provided with a manual switch to stop treatment any time. Preset lumbar disc herniation protocol was used. Each session lasted fifteen minutes, applied force had 100-gram step increments, and did not exceed 50% of the weight of the patient. At the end of the therapy, the cord was disconnected and belts were removed. Participants were asked to sit for three minutes to identify any adverse reaction.

SUMMARY:
The goal of this quasi-experimental trial was to evaluate the effects of non-surgical spinal decompression on disability and pain in patients with chronic low back pain and sciatica throughout a two-month follow-up, and to analyze the relationship between demographic factors and clinical outcomes after a program of non-surgical spinal decompression.

The main questions it aims to answer were:

* Non-surgical spinal decompression is effective to reduce pain intensity and self-reported disability in patients with chronic low back pain and sciatica?
* Age, level of education and work activities are related with clinical outcome in patients treated with non-surgical spinal decompression?

Participants underwent eight sessions, three per week, with the BTL-6000 spinal decompression system. The study did not have a comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years old.
* Chronic (at least six months) low back pain (LBP) and/or sciatica.
* Abnormalities of intervertebral disc on magnetic resonance imaging (MRI).

Exclusion Criteria:

* Patients with prior spine surgery.
* Vertebral instability.
* Cancer.
* Current infectious disease.
* Pregnancy.
* Kinesiophobia.
* Fibromyalgia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Self-reported disability | Baseline, at the end of the eighth session, and at 2nd-month follow-up.
  We measured self-reported disability associated with spine disorders through the spanish version of the Oswestry Disability Index (ODI), a reliable and validated instrument composed by ten sections (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and traveling), in which the patient grades the disability from zero (no limitation) to five (limitation prevents me from performing the activity). The ODI final score was calculated with the following formula: [total score/(5 x number of answered questions)] x 100%, and interpreted as the higher the score, the greater the disability.
Pain intensity | Baseline, at the end of the eighth session, and at 2nd-month follow-up.
  Pain intensity was also evaluated with the numeric pain rating scale (NPRS), a popular clinical tool consisting of a numbered straight line from zero (no pain) to ten (the worst pain), where the patients registered their current pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Tonatiuh Avila, MD, Principal Investigator — Hospital Civil de Guadalajara
Locations (1):
- Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author, upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: No determined.